CLINICAL TRIAL: NCT04793464
Title: Scaling Up SARS-CoV-2 Testing to Serve Latinx Communities
Brief Title: COVID-19: Healthy Oregon (Oregon Saludable): Together We Can (Juntos Podemos)
Acronym: OSJP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Leslie Leve,, Lorry Lokey Professor, College of Education; Associate Director, Prevention Science Institute, University of Oregon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10032020.002; P50DA048756-02S2 (NIH)
Record Dates: First submitted 2021-02-25; First posted 2021-03-11 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Health Behavior; Health Care Utilization
Keywords: Latinx; SARS-CoV-2; COVID-19; Hispanic; Testing
MeSH Terms: conditions — Health Behavior; Patient Acceptance of Health Care; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Promotores (Experimental): The Promotores de Salud intervention involves specified outreach and psychoeducation on SARS-CoV-2 health related behaviors.
  Interventions: Behavioral: Promotores de Salud
- Control (Active Comparator): Services as usual includes outreach as usual strategies and pamphlets on site at events.
  Interventions: Behavioral: Services as usual

INTERVENTIONS:
Behavioral: Promotores de Salud — The Promotores de Salud intervention is delivered by a paid Promotor(a) who is a trusted member of the community where the testing site is located. The intervention includes: (1) psychoeducation to increase knowledge about COVID-19 and the benefits of testing; (2) motivational interviewing (MI) strategies to explore personal, social, and behavioral barriers to testing and to discuss available resources to resolve these barriers; (3) emotional support to address testing-related concerns and anxieties that may dissuade Latinx individuals from getting tested; and (4) service navigation. When promotores are on-site at testing events, they will provide information about COVID-19 and preventive behaviors using in-person instruction on effective mask wearing, hand washing, and physical distancing, as well as the importance of repeated testing and vaccines.
  Other Names: Promotores
  Arms: Promotores
Behavioral: Services as usual — Services as usual, our control condition, includes strategies that are typically conducted by county and community-based organizations that serve under-represented groups to notify people of testing opportunities related to COVID-19. These include Facebook advertisements, email announcements, circulation to other community-based organizations and state agencies (e.g., Oregon Health Authority, county public health), and other flyer distribution means. This condition also includes a pamphlet about health behaviors and community resources handed out by testing facilitators at testing events.
  Other Names: Control
  Arms: Control

SUMMARY:
The global SARS-CoV-2 pandemic that causes the severe respiratory illness COVID-19 is the worst health crisis that the United States has faced in a century. Although this highly contagious virus has infected millions of Americans already, the disease burdens are disproportionately born by historically underserved populations such as Latinx communities. This disparity is notable in Oregon, where the 13% of the population that is Latinx represents approximately 44% of COVID-19 cases. An urgent need exists to reach Oregon's Latinx community to prevent SARS-CoV-2 transmission.

The overall goal of this study is to implement a Promotores de Salud intervention to increase the reach, access, uptake, and impact of testing in Latinx communities in Oregon. This project will fully integrate with the National institutes of Health (NIH) Rapid Acceleration of Diagnostics (RADx) consortium and its Coordination and Data Collection Center (CDCC). With guidance and leadership from the study's Latinx Community and Scientific Advisory Board, 38 testing sites have been established to test the Promotores de Salud intervention. The investigators will test whether the Promotores de Salud intervention will increase testing rates and promote better health behaviors in communities over time. The investigators will test the intervention using a randomized control trial comparing the intervention to county outreach services as usual. Evaluation of the Promotores de Salud intervention held during a testing event (compared to distribution of a pamphlet only) will test whether culturally competent education results in greater use of strategies that reduce transmission of COVID-19 at the community and individual level.

The investigators have designed a working group structure with teams focused on: Community Engagement, Molecular Biology, Data Science, and Implementation Science. These working groups are coordinated by an Administrative Hub and guided by the study's Latinx Community and Scientific Advisory Board.

Over time, this project will help communities institutionalize optimal local testing frameworks supported by University of Oregon laboratory facilities for testing capacity, technical support for testing logistics, and collection of data on health behaviors, testing rates, and sustainability. The resulting structures and systems will be poised for future scale-up to other vulnerable communities and/or for other public health purposes (e.g., vaccination campaigns).

DETAILED DESCRIPTION:
A total of 38 communities have established a testing site with testing events held every other week (bi-weekly). The study randomized counties at the site level within county. The investigators used a priori stratification by county as sample size is small. Half of all sites in a county were assigned to the control condition (services as usual), and the other half to the intervention condition (Promotores de Salud). Randomly assigned communities receive one of two outreach strategies: Services as usual (culturally tailored flyers, radio announcements, social media posts, health behavior pamphlet on site) or services as usual plus the Promotores de Salud intervention, where a paid, trusted community member reaches out to community members to motivate them to utilize the free testing services and improve COVID-19 related health behaviors. The Promotores de Salud intervention was designed to build relationships with Latinx community members and facilitate trust.

To assess the proportion of Latinx community members tested at each site, the investigators will use de-identified health information provided to the study by the University of Oregon's (UO) COVID-19 clinical genomics laboratory, who are processing the tests. To assess health behaviors, a subset of adult participants at each site will be invited to participate in a research survey, administered at baseline and again 30 days later. For both approaches, the study anticipates engaging a greater proportion Latinx community members, relative to overall county demographics. The overall study population is expected to be 85% Hispanic and 15% non-Hispanic, with 84% of individuals identifying as White in both ethnic groups and the remaining 16% identifying as African American, Asian, Pacific Islander, American Indian/Alaska Native, or more than one race. There will be 19 sites per study group (38 total) and up to roughly 3,600 adult individuals in the intervention (n = 1,800) or control conditions (n = 1,800).

This study also leverages data from a patient registry from the University of Oregon's COVID-19 clinical genomics laboratory.

Quality Assurance, Data Checks, Source Data Verification, Data Dictionary, and Standard Operating Procedures: Data and biospecimens will be collected in-person at testing sites, requiring direct interaction with participants. In order to report SARS-CoV-2 infection results back to each participant, name, date of birth, and contact information are collected. To fulfill reporting requirements to the Oregon Health Authority, county of residence and zip code are also collected for each person tested. Data used to evaluate the efficacy of intervention will involve aggregate variables derived from data collected as part of the diagnostic testing procedure and will be aggregated at the level of the testing site (e.g., tests performed, race and ethnicity percentages, etc.).

For the collection of SARS-CoV-2 samples, testing facilitators will guide participants in the self-collection process. For anterior nares, participants are instructed to place the nasal swab about 1cm into their nostril and rotate it, making contact with the nasal membrane for 10 seconds, then repeating the process with the same swab in the other nostril. Parents are instructed to collect the sample for their child if the child is under 10 years old, or if the minor child requests parental assistance. Testing site staff can assist participants who have low dexterity or physical impairments in sample collection. In case of an injury during sample collection, the partnering community organization staff will direct the participant to the appropriate medical resources. Samples will be placed into sterile barcoded vials (1 ml Matrix, barcoded screw-cap tubes) that each contain 500 microliters (μl) of DNA/RNA Shield. Each Matrix tube will then be closed tightly and will be placed in a standard plastic laboratory microcentrifuge tube rack with eight rows and twelve columns (8-by-12 rack with 96 positions). This rack will then be externally decontaminated by brief submersion in accelerated hydrogen peroxide (H202). Each 96-position microcentrifuge tube rack will then be labeled and placed in a sterile temporary container with wet ice at 4Cdegrees. If possible at each site, racks will be periodically transferred either to a refrigerator (4C) or freezer (-20C) for storage. At the end of the day all racks will be transported on wet ice to the COVID-19 clinical genomics Laboratory at UO, ensuring that they will arrive no longer than 48 hours after collection and preferably within 12-24 hours. If the testing site is located too distally for hand transport, tube racks will be secured and shipped by express methods on dry ice.

Each 96 well collection plate will next proceed to molecular processing using the standard, FDA approved Thermo Fisher TaqPath analysis protocol. All steps of this approved protocol will be followed exactly, including the appropriate reagents, volumes, and inclusion of appropriate positive and negative controls. In addition, investigators will employ the software analysis system and parameters exactly as specified. First, RNA will be extracted from each well using the MagMax Viral/Pathogen Nucleic Acid Isolation Kit (ThermoFisher, #100081242) which removes potentially inhibiting contamination and increases the sensitivity and consistency of subsequent qPCR protocols. Depending upon the number of samples to be processed, the RNA extraction will either occur by hand using multichannel pipettors or through the use of the Hamilton Robot. The purified RNA will then be retrotranscribed for analysis using the TaqPath RT-PCR COVID-19 Kit on either 96 well or 384 well QuantStudio5 (QS5) thermocyclers depending upon the number of samples to be processed. If the lab technicians need to process 384 samples, they will use the Hamilton liquid handling robot (Hamilton, Microlab VANTAGE 2.0) to aliquot from each of four-96 well plates into the 384 well plate format for subsequent qPCR amplification. In this RT-PCR process, probes anneal to three unique forward and reverse primers for three SARS-CoV-2 genes: ORF1ab, N Protein and S Protein.

All laboratory and reporting will be automated through the use of barcodes, robotics, 96 and 384 well qPCR machines, and the use of a fully HIPAA and CAP3 compliant Laboratory Information Management System (LIMS) built by L7 informatics (https://l7informatics.com/). These system automations and use of LIMS allow increased throughput (up to several thousand samples per day) and rapid analysis and automated reporting of results through the LIMS. The qPCR data are stored in the LIMS system for analysis using the Applied Biosystems COVID-19 Interpretive Software to allow a qualitative assessment of whether the virus is present in the sample (a 'positive' case), absent, or uncertain. The LIMS system in the COVID-19-MAP lab allows the integration of this analysis software into the appropriate step of the overall sample tracking workflow pipeline, and therefore the immediate result can be linked to the appropriate barcode in the database. Furthermore, the LIMS system is connected and communicates via a local area network (LAN) with all equipment (e.g., robots and qPCR machines) to document each step of the process for CLIA validation. The results for each sample, and associated metadata on the steps during processing, are then associated with each assigned barcode and can then be disseminated, as appropriate, to the Oregon Health Authority, the appropriate county health department, and the individual. Test results will be available within 48 hours and no later than 4 days to the individual and/or the health authority.

After testing occurs, researchers will have access to aggregate, community-level (e.g., counts and prevalence rates), de-identified data prepared by the UO's CLIA clinical genomics laboratory. The data will include four protected health identifiers: site zip code, participant zip code, testing result, and testing date. It will also include demographic data this is not protected health information such as age range, race, and ethnicity. These data will be used to assess outreach activities aimed at increasing participation of Latinx community members in SARS-COV-2 testing. The primary outcome for this aspect of the study is site-level testing rates of Latinx individuals.

Sample Size Assessment, Plan for Missing Data, Statistical Analysis Plan: For the primary efficacy evaluation of the Promotores intervention, the investigators will employ standard normal theory analysis of covariance (ANCOVA) and auto-regressive linear modeling for continuous outcomes such as COVID-19 knowledge; and they will employ pre-post generalized linear modeling for count and ordered categorical outcomes such as proportion of Latinx tested at each geographic site. To address the non-independence of participants in the intervention design, investigators will estimate linear mixed models. Two primary sources of missing data are expected, item non-response and attrition over time. For dropout, investigators will conduct standard attrition analyses to compare baseline characteristics between attriters and completers. They will consider propensity score matching procedures and complier average causal effects models to address substantial differences. For item non-response and scale score development, investigators will require 70% of scale items be present for scoring. They will test whether scale level data are missing completely at random (MCAR) within waves and then across waves. If data are not MCAR, under assumptions of missing at random (MAR, i.e., data are not dependent on missing values of the intervention response variable), investigators will employ one of two recommended approaches for SEM, full information maximum likelihood (FIML) or multiple imputation (MI). Although these approaches can be problematic when data are non-ignorable missing, they are still recommended for handling missingness, particularly with covariates associated with attrition. Both methods provide more efficient standard errors than listwise or pairwise deletion, or mean substitution. Should missing data or attrition be associated with covariates, investigators will include appropriate covariates in hypothesis testing. For the pre-post individual level criterion outcomes, 38 sites with roughly 50 to 100 participants per site plus attrition (n = 2160) an alpha level of .05 and intra-class correlations ranging from .05 to .20 provides power to detect effects ranging from .19 to .32, respectively (small to moderate).

Finally, data will be collected in accordance with Tier 1 "common data elements" from the national Duke Coordination and Data Collection Center (CDCC). The CDCC directly assists each individual RADx-UP project to optimize engagement, outreach, testing strategies, and to facilitate co-learning opportunities between and among RADx-UP projects. Key outcome data and the testing procedures for obtaining the sample, analysis platform, analysis procedures, and test resulting will be collected and represented in a consistent manner for harmonization across the consortium, integrated with test reporting requirements under the Coronavirus Aid, Relief, and Economic Security Act (CARES Act).

ELIGIBILITY:
Inclusion Criteria:

* Proportion Tested: Age 3 or older
* Proportion Tested: Received testing at study testing site
* Individual Survey: 15 or older

Exclusion Criteria:

• Individual Survey: Unable to understand Spanish or English or another language translated by a qualified translator at a 5th grade level

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1623 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie D Leve, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share IPD with the RADx-Up CDCC. All Tier 1 data elements required by the CDCC will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be shared in accordance with timeframes set by the RADX-UP CDCC
Access Criteria: The RADX-UP CDCC will make these determinations
URL: https://radx-up.org/about/

REFERENCES:
- [Background] Budd EL, McWhirter EH, De Anda S, Mauricio AM, Mueller MV, Cioffi CC, Nash A, Van Brocklin K, Yarris K, Jackson A, Terral H, Ramirez Garcia JI; Juntos Podemos Community and Scientific Advisory Board; Cresko WA, DeGarmo DS, Leve LD. Development and design of a culturally tailored intervention to address COVID-19 disparities among Oregon's Latinx communities: A community case study. Front Public Health. 2022 Sep 23;10:962862. doi: 10.3389/fpubh.2022.962862. eCollection 2022. PMID 36211681
- [Result] Searcy JA, Cioffi CC, Tavalire HF, Budd EL, Cresko WA, DeGarmo DS, Leve LD. Reaching Latinx Communities with Algorithmic Optimization for SARS-CoV-2 Testing Locations. Prev Sci. 2023 Aug;24(6):1249-1260. doi: 10.1007/s11121-022-01478-x. Epub 2023 Jan 9. PMID 36622480
- [Result] Anda S, Budd EL, Halvorson S, Mauricio AM, McWhirter EH, Cioffi CC, Garcia JIR, Cresko WA, Leve LD, DeGarmo DS. Effects of a Health Education Intervention for COVID-19 Prevention in Latinx Communities: A Cluster-Randomized Controlled Trial. Am J Public Health. 2022 Nov;112(S9):S923-S927. doi: 10.2105/AJPH.2022.307129. PMID 36446063
- [Result] DeGarmo DS, De Anda S, Cioffi CC, Tavalire HF, Searcy JA, Budd EL, Hawley McWhirter E, Mauricio AM, Halvorson S, Beck EA, Fernandes L, Currey MC, Ramirez Garcia J, Cresko WA, Leve LD. Effectiveness of a COVID-19 Testing Outreach Intervention for Latinx Communities: A Cluster Randomized Trial. JAMA Netw Open. 2022 Jun 1;5(6):e2216796. doi: 10.1001/jamanetworkopen.2022.16796. PMID 35708690
- [Derived] Ramirez Garcia JI, Oro V, Budd EL, Mauricio AM, Cioffi CC, Anda S, McWhirter EH, DeGarmo DS, Leve LD. A Translational Case Study of a Multisite COVID-19 Public Health Intervention Across Sequenced Research Trials: Embedding Implementation in a Community Engagement Phased Framework. Am J Public Health. 2024 May;114(S5):S396-S401. doi: 10.2105/AJPH.2024.307669. PMID 38776498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initial recruitment occurred at the testing sites. A standardized recruitment script was used and will include eligibility questions including: (1) age, (2) attendance at event, (3) able to understand English or Spanish at a 5th grade level, (4) was not previously enrolled in the project. Re-recruitment occurred 30 days after enrollment. Participants were asked in the first survey how they preferred to complete the follow-up survey, with options to complete by phone, mail, or online.
Groups:
- Unknown Treatment Status: Exposure status unknown, but data collected
Period: Overall Study
Arm/Group | Promotores | Control | Unknown Treatment Status
Started (Enrolled at Baseline) | 1125 | 483 | 15
Completed (Completed Follow-up) | 624 | 300 | 10
Not Completed | 501 | 183 | 5
Not completed — Lost to Follow-up | 458 | 168 | 5
Not completed — Withdrawal by Subject | 43 | 15 | 0

BASELINE CHARACTERISTICS:
Population: 1623 participants were recruited at baseline. Of those 1623, 1125 were assigned to a site of the intervention condition, 483 were assigned to a site of the control condition, 15 completed the BL enrollment, but their site identifiers were missing.
Groups:
- Total: Total of all reporting groups
Arm/Group | Promotores | Control | Unknown Treatment Status | Total
Number analyzed (Participants) | 1125 | 483 | 15 | 1623
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (15.7) | 39.0 (14.4) | 35.4 (14.0) | 40.4 (15.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Male | 440 | 188 | 5 | 633
  Sex/Gender: Female | 647 | 288 | 8 | 943
  Sex/Gender: Unknown | 38 | 7 | 2 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 776 | 325 | 6 | 1107
  Not Hispanic or Latino | 302 | 151 | 6 | 459
  Unknown or Not Reported | 47 | 7 | 3 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 120 | 63 | 3 | 186
  Asian | 17 | 12 | 0 | 29
  Native Hawaiian or Other Pacific Islander | 4 | 6 | 0 | 10
  Black or African American | 7 | 9 | 0 | 16
  White | 280 | 136 | 7 | 423
  More than one race | 36 | 23 | 0 | 59
  Unknown or Not Reported | 661 | 234 | 5 | 900
Region of Enrollment [Number; unit: participants]
  United States | 1125 | 483 | 15 | 1623
COVID-19 Prevention Health Behaviors 1 [Mean (Standard Deviation); unit: units on a scale] — From the PhenX toolkit, Protocol - COVID-19 Knowledge, Attitudes, and Avoidant Behaviors, participants are asked to indicate "Which of the following have you done in the last seven days to keep yourself safe from coronavirus? Only consider actions that you took or decisions that you made personally." There are a total of 17 possible items participants rate as a binary, Yes/No, response. The count of 'yes' responses was recorded. The scale will range from 0-17. A higher score indicates more preventative behaviors.
  units on a scale | 6.2 (3.8) | 7.4 (4.0) | 7.0 (4.7) | 6.6 (3.9)
COVID-19 Prevention Health Behaviors 2 [Mean (Standard Deviation); unit: units on a scale] — From the PhenX toolkit, Protocol - COVID-19 Knowledge, Attitudes, and Avoidant Behaviors, participants are asked to indicate "Which of the following have you done in the last five days?" There are 5 items that increase risk for COVID-19, rated on a checklist (check indicates participation in behavior). A mean was taken across all items. The scale ranges from 0-5 with 5 indicating greater risk behavior.
  units on a scale | 1.3 (1.5) | 1.4 (1.4) | 1.4 (1.0) | 1.3 (1.5)
COVID-19 Knowledge and Attitudes 1 [Count of Participants; unit: Participants] — Participants are asked, "How can the novel coronavirus be transmitted?" adapted from the PhenX toolkit COVID-19 COMMUNITY RESPONSE SURVEY, KNOWLEDGE & ATTITUDES TOWARDS COVID-19. Participants to indicate using a Yes/No response to 'Close contact with an infected person who has symptoms'. Counts of 'yes' responses are given. Population: Not all participants responded to this item.
  Participants
    number analyzed (Participants) | 719 | 383 | 10 | 1112
    (all) | 624 | 317 | 10 | 951
COVID-19 Knowledge and Attitudes 2 [Count of Participants; unit: Participants] — Participants are asked, "How can the novel coronavirus be transmitted?" adapted from the PhenX toolkit COVID-19 COMMUNITY RESPONSE SURVEY, KNOWLEDGE & ATTITUDES TOWARDS COVID-19. Participants to indicate using a Yes/No response to "Close contact with an infected person even if they aren't showing symptoms of infection". Counts of 'yes' responses are provided. Population: Not all participants responded to this item.
  Participants
    number analyzed (Participants) | 715 | 386 | 11 | 1112
    (all) | 627 | 315 | 11 | 953
COVID-19 Knowledge and Attitudes 3 [Mean (Standard Deviation); unit: units on a scale] — Participants were asked: "In your opinion, how effective are the following actions for keeping you safe from COVID-19?" A list of 6 prevention strategies are listed. Participants indicate their response on a scale Very Effective (5) to Not Effective at All (1). A mean score is computed. A higher score indicates a preferable outcome. Population: Not all participants responded to this item.
  units on a scale
    number analyzed (Participants) | 750 | 407 | 12 | 1169
    (all) | 4.2 (0.8) | 4.2 (0.8) | 4.4 (0.7) | 4.2 (0.8)
COVID-19 Knowledge and Attitudes 4 [Mean (Standard Deviation); unit: units on a scale] — Participants were asked: "How safe or unsafe are the following actions for avoiding exposure to coronavirus?" A list of 11 activities are listed and responses are on scale of 1 (Extremely Unsafe) to 4 (Extremely Safe). Mean score was calculated. Lower scores indicate less caution. Population: Not all participants responded to this item.
  units on a scale
    number analyzed (Participants) | 724 | 393 | 12 | 1129
    (all) | 2.4 (0.6) | 2.4 (0.6) | 2.6 (0.4) | 2.4 (0.6)
Attitudes Towards COVID-19 Vaccines [Mean (Standard Deviation); unit: units on a scale] — Participants are asked, "How likely are you to get vaccinated for coronavirus once a vaccination is available to the public?" on a 5-item response scale of "Very likely" to "Definitely not". The mean of these items will be computed on a scale of 1-5 with 5 indicating greater likelihood of receiving the vaccine and lower vaccine hesitancy. Population: Not all participants responded to this item.
  units on a scale
    number analyzed (Participants) | 699 | 330 | 10 | 1039
    (all) | 4.6 (0.9) | 4.6 (0.9) | 4.7 (0.7) | 4.6 (0.9)
Broadband Internalizing Symptoms [Mean (Standard Deviation); unit: units on a scale] — Participants respond to the Phenx Toolkit depression (2 items) and anxiety (2 items) subscales regarding how much or how often they have been bothered by each problem during the past 2 weeks. Items are rated on a scale ranging from 0-4, where 0="none/not at all" and 4= "severe/nearly every day". A mean score will be computed from the 4 items, with higher scores indicating more symptoms. Population: Not all participants responded to this item.
  units on a scale
    number analyzed (Participants) | 1053 | 459 | 12 | 1524
    (all) | 1.6 (0.9) | 1.7 (1.0) | 2.0 (1.1) | 1.7 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Prevention Health Behaviors 1
Description: From the PhenX toolkit, Protocol - COVID-19 Knowledge, Attitudes, and Avoidant Behaviors, participants are asked to indicate "Which of the following have you done in the last even days to keep yourself safe from coronavirus? Only consider actions that you took or decisions that you made personally." There are a total of 17 possible items participants rate as a binary, Yes/No, response. The count of 'yes' responses was recorded. The scale will range from 0-17. A higher score indicates more preventative behaviors.
Time Frame: Change from baseline health behaviors at 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promotores | Control | Unknown Treatment Status
Number analyzed (Participants) | 624 | 300 | 10
score on a scale | 6.0 (3.6) | 6.7 (3.9) | 4.8 (2.6)
Statistical Analysis 1: Comparison: Promotores vs Control; Number analyzed is the number of participants with valid baseline and follow-up data; Test type: Superiority; p = .26, ANCOVA; Mean Difference (Final Values) = .77

2. Primary Outcome: COVID-19 Prevention Health Behaviors 2
Description: From the PhenX toolkit, Protocol - COVID-19 Knowledge, Attitudes, and Avoidant Behaviors, participants are asked to indicate "Which of the following have you done in the last five days?" There are 5 items that increase risk for COVID-19, rated on a checklist (check indicates participation in behavior). A mean was taken across all items.The scale ranges from 0-5 with 5 indicating greater risk behavior.
Time Frame: Change from baseline health behaviors at 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promotores | Control | Unknown Treatment Status
Number analyzed (Participants) | 624 | 300 | 10
score on a scale | 1.4 (1.5) | 1.7 (1.5) | 2.1 (1.7)
Statistical Analysis 1: Comparison: Promotores vs Control; Number analyzed is the number of participants with valid baseline and follow-up data; Test type: Superiority; p = .02, ANCOVA; Ratio of Means; Mean Difference (Final Values) = .87

3. Primary Outcome: COVID-19 Knowledge and Attitudes 1
Description: Participants are asked, "How can the novel coronavirus be transmitted?" adapted from the PhenX toolkit COVID-19 COMMUNITY RESPONSE SURVEY, KNOWLEDGE & ATTITUDES TOWARDS COVID-19. Participants to indicate using a Yes/No response to "Close contact with an infected person who has symptoms". Counts of 'yes' responses are given.
Time Frame: Change from baseline COVID-19 attitudes and knowledge at 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Promotores | Control | Unknown Treatment Status
Number analyzed (Participants) | 380 | 224 | 6
Participants | 325 | 187 | 5
Statistical Analysis 1: Comparison: Promotores vs Control; Number analyzed is the number of participants with valid baseline and follow-up data; Test type: Superiority; p = .68, ANCOVA; Logistic regression; Odds Ratio (OR) = 1.10

4. Primary Outcome: COVID-19 Knowledge and Attitudes 2
Description: Participants are asked, "How can the novel coronavirus be transmitted?" adapted from the PhenX toolkit COVID-19 COMMUNITY RESPONSE SURVEY, KNOWLEDGE & ATTITUDES TOWARDS COVID-19. Participants to indicate using a Yes/No response to 'Close contact with an infected person even if they aren't showing symptoms of infection'. Counts of 'yes' responses are provided.
Time Frame: Change from baseline COVID-19 attitudes and knowledge at 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Promotores | Control | Unknown Treatment Status
Number analyzed (Participants) | 391 | 228 | 7
Participants | 335 | 187 | 6
Statistical Analysis 1: Comparison: Promotores vs Control; Number analyzed is the number of participants with valid baseline and follow-up data; Test type: Superiority; p = .44, ANCOVA; Logistic regression; Odds Ratio (OR) = 1.19

5. Primary Outcome: COVID-19 Knowledge and Attitudes 3
Description: Participants were asked: "In your opinion, how effective are the following actions for keeping you safe from COVID-19?" A list of 6 prevention strategies are listed. Participants indicate their response on a scale Very Effective (5) to Not Effective at AlI (1). Scale range is 1-5. A mean value is computed. Higher scores indicate a better outcome.
Time Frame: Change from baseline COVID-19 attitudes and knowledge at 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promotores | Control | Unknown Treatment Status
Number analyzed (Participants) | 409 | 239 | 7
score on a scale | 4.1 (0.7) | 4.1 (0.8) | 4.2 (0.6)
Statistical Analysis 1: Comparison: Promotores vs Control; Number analyzed is the number of participants with valid baseline and follow-up data; Test type: Superiority; p = .77, ANCOVA; Mean Difference (Final Values) = .015

6. Primary Outcome: COVID-19 Knowledge and Attitudes 4
Description: Participants were asked: "How safe or unsafe are the following actions for avoiding exposure to coronavirus?" A list of 11 activities are listed and responses are on scale of 1 (Extremely Unsafe) to 4 (Extremely Safe). Mean scores were calculated. Scores range between 1-4. Higher score means a worse outcome.
Time Frame: Change from baseline COVID-19 attitudes and knowledge at 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promotores | Control | Unknown Treatment Status
Number analyzed (Participants) | 389 | 234 | 7
score on a scale | 2.5 (0.5) | 2.4 (0.5) | 2.6 (0.2)
Statistical Analysis 1: Comparison: Promotores vs Control; Number analyzed is the number of participants with valid baseline and follow-up data; Test type: Superiority; p = .66, ANCOVA; Mean Difference (Final Values) = .017

7. Primary Outcome: Attitudes Towards COVID-19 Vaccines
Description: Participants are asked, "How likely are you to get vaccinated for coronavirus once a vaccination is available to the public?" on a 5-item response scale of "Very likely" to "Definitely not". The item was computed on a scale of 1-5 with 5 indicating greater likelihood of receiving the vaccine and lower vaccine hesitancy. Higher scores indicate a better outcome.
Time Frame: Change from baseline attitudes towards COVID-19 vaccines at 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promotores | Control | Unknown Treatment Status
Number analyzed (Participants) | 323 | 172 | 7
score on a scale | 4.6 (0.9) | 4.6 (1.0) | 4.7 (0.5)
Statistical Analysis 1: Comparison: Promotores vs Control; Number analyzed is the number of participants with valid baseline and follow-up data; Test type: Superiority; p = .44, ANCOVA; Mean Difference (Final Values) = -.05

8. Secondary Outcome: Broadband Internalizing Symptoms
Description: Participants respond to the Phenx Toolkit depression (2 items) and anxiety (2 items) subscales regarding how much or how often they have been bothered by each problem during the past 2 weeks. Items are rated on a scale ranging from 0-4, where 0="none/not at all" and 4= "severe/nearly every day". A mean score will be computed from the 4 items, with higher scores indicating more symptoms. Higher scores indicate a worse outcome.
Time Frame: Change from baseline symptoms at 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promotores | Control | Unknown Treatment Status
Number analyzed (Participants) | 577 | 281 | 8
score on a scale | 1.7 (0.8) | 1.9 (1.0) | 1.6 (0.7)
Statistical Analysis 1: Comparison: Promotores vs Control; Number analyzed is the number of participants with valid baseline and follow-up data; Test type: Superiority; p = 0.017, ANCOVA; Mean Difference (Final Values) = -.12

ADVERSE EVENTS:
Time Frame: No adverse event data reported. Adverse events were monitored/assessed through study completion, approximately 6 months.
Arm/Group | Promotores | Control | Unknown Treatment Status
All-Cause Mortality (participants affected / at risk) | 0/1125 | 0/483 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/1125 | 0/483 | 0/15
Other Adverse Events (participants affected / at risk) | 0/1125 | 0/483 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT04793464/Prot_001.pdf
  • Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT04793464/SAP_002.pdf
  • Informed Consent Form (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT04793464/ICF_000.pdf